CLINICAL TRIAL: NCT00609934
Title: A Phase I/II Study of Sorafenib and Palliative Radiotherapy in Patients With Advanced Renal Cell Carcinoma and Symptomatic Bony Metastases
Brief Title: Study of Sorafenib and Palliative Radiotherapy in Kidney Cancer That Spreads to the Bone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DDPDRO-004; UHN REB 07-0357-C
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Renal Cell Carcinoma
Keywords: renal cell carcinoma; kidney cancer; bone metastases; RCC; bone pain; palliative radiotherapy; sorafenib; radiation; renal cell
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib and palliative radiotherapy (Experimental)
  Interventions: Drug: Sorafenib; Radiation: external beam radiotherapy

INTERVENTIONS:
Drug: Sorafenib — Dose level 1: sorafenib 200mg PO OD on Days 1-84 Dose level 2: sorafenib 400mg PO OD on Days 1-84
  Other Names: BAY 43-9006; NSC 724772
Radiation: external beam radiotherapy — 3000cGy in 10 fractions

SUMMARY:
The purpose of this study is to investigate the use of a new anti-angiogenic drug called sorafenib, in combination with radiotherapy, for renal cell cancer that has spread to the bone and is causing significant pain. The study will find a safe dose of sorafenib for this combination study treatment, look at side effects, and test if the study treatment is effective in controlling the pain experienced from this type of renal cell cancer. . There will be two parts or phases to this study

The purpose of the first phase is to find the highest dose of sorafenib that can be given safely to patients, when combined with radiotherapy. We will also see what kind of effects the study treatment has on you and your cancer. Participants in this phase will receive a dose of sorafenib that has shown to be well-tolerated in humans. If the side effects are tolerable for this dose of sorafenib when combined with radiotherapy, new patients will be asked to join the study and will receive a dose of sorafenib higher than the last study participant.

In the second phase, new study participants will receive the dose of sorafenib that was determined to be safe in the first phase. Side effects will continue to be looked at and the effectiveness on controlling pain symptoms from this type of cancer, will also be looked at.

ELIGIBILITY:
Eligibility Criteria

1. Eligible patients must have histologically or cytologically confirmed metastatic RCC that is judged to be incurable with standard therapy.
2. Patients must have at least one radiographically-evident symptomatic (> 2/10 on the Brief Pain Inventory) bone metastasis that is amenable to palliative radiation. Multiple symptomatic bone metastases may be irradiated at the same time. However, if more than one symptomatic bone metastasis is identified, one will be chosen as the index lesion for reporting purposes.
3. No planned change in analgesic medications.
4. No planned increase in regular analgesic medications.
5. No prior surgery to the index lesion, although previous surgery for other metastatic disease is permissible if > 4 weeks prior to study registration.
6. Patients may have had up to two previous lines of systemic treatment for metastatic RCC, including prior treatment with sorafenib or another similar multi-targeted tyrosine kinase inhibitor, if completed >4 weeks prior to study registration.
7. Patients may not have had previous radiotherapy to the index lesion. Patients may have had previous radiotherapy to other metastases if completed > 4 weeks prior to study registration. Patients must have recovered from the acute side effects of radiotherapy prior to study registration.
8. Age >18 years.
9. Life expectancy of greater than 3 months.
10. ECOG performance status < 2 (Karnofsky > 60).
11. Patients must have normal organ and marrow function as defined below:

    i. Absolute neutrophil count >1.5 x109 /L ii. Platelet count >75 x109 /L iii. Total bilirubin < 1.5 x ULN iv. AST (SGOT) / ALT (SGPT) < 2.5 × institutional ULN or < 5 x institutional ULN if liver metastases v. Creatinine <1.7 x ULN or vi. Creatinine clearance > 50 mL/min/1.73 m2 vii. International Normalized Ratio (INR) < 1.5 viii. Hemoglobin value Hb > 80 g/L ix. Serum phosphate level > 0.80 mmol/L x. Serum lipase, normal values (range of 5-208 U/L) xi. Serum amylase, normal values (range 30-110 U/L)
12. Ability to understand and the willingness to sign a written informed consent document.
13. The effects of sorafenib on the developing human fetus at the recommended therapeutic dose are unknown. Women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation. Effective methods of birth control would include a barrier method (e.g. condoms, diaphragm) combined with spermicide, or an intrauterine device (IUD). Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria

1. Serious medical condition that might be aggravated by treatment, including but not limited to: myocardial infarction within 6 months, congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, uncontrolled hypertension, uncontrolled psychotic disorders, serious infections, active peptic ulcer disease, active liver disease, or cerebrovascular disease with previous stroke.
2. Patients may not be receiving any other investigational agent concurrently or within 4 weeks of study registration. Patients receiving other molecularly-targeted treatments for RCC off of study, including inhibitors of angiogenesis or mTOR, will be eligible for this study after a 1 week wash-out period.
3. Patients with clinical or radiological evidence of spinal cord compression are ineligible.
4. Patients who are at high risk of pathologic fracture and appropriate for surgical intervention are ineligible.
5. Patients who are planned for palliative surgical intervention to the index lesion or adjacent bone are ineligible.
6. Pregnant or lactating women are excluded from this study because the safety of sorafenib has not been established in these circumstances.
7. Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with sorafenib.
8. Patients with other active malignancies other than non-melanoma skin cancer are excluded.
9. Patients who have had significant surgical procedures requiring a general anaesthetic (for example, open laparotomy or thoracotomy) within the past month
10. Patients who possess significant unhealed wounds or ulcers
11. Patients with any bleeding or clotting disorder
12. Patient taking greater than 325mg of aspirin per day
13. Patients with diabetes mellitus will be ineligible for the PET-CT components of the study, but will remain eligible to receive sorafenib.
14. Patients who are currently taking rifampin, phenytoin, carbamazepine, Phenobarbital, dexamethasone and St. John's Wort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Reduction in pain from index lesion 4 weeks following the completion of radiotherapy, assessed using Brief Pain Inventory. | 7 weeks

SECONDARY OUTCOMES:
reduction in pain in index lesion at study termination assessed using Brief Pain Inventory | 12 weeks
acute toxicity of palliative radiotherapy and sorafenib together | 12 weeks
acute toxicity of sorafenib alone | 1 week
biologic response of the index lesion to radiotherapy and sorafenib assessed using FDG-PET-CT | 7 weeks
disease-free survival | greater than 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hosptial, Toronto, Ontario, Canada